CLINICAL TRIAL: NCT01255800
Title: A Pilot Study of Cetuximab and the Hedgehog Inhibitor IPI-926 in Recurrent Head and Neck Cancer: a Rational Anti-Cancer Stem Cell Combination.
Brief Title: Pilot Study of Cetuximab and the Hedgehog Inhibitor IPI-926 in Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0109.cc
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Recurrent Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — IPI-926; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IPI-926 and Cetuximab (Experimental): * Patients will receive Cetuximab IV every week.
  * Starting on Day 15 of the first cycle, Patients will take the study drug by mouth every day.
  Interventions: Drug: IPI-926 and Cetuximab

INTERVENTIONS:
Drug: IPI-926 and Cetuximab — * Patients will receive Cetuximab IV every week.
  * Starting on Day 15 of the first cycle, Patients will take IPI-926by mouth every day.
  Other Names: brand name: ERBITUX

SUMMARY:
This study will evaluate the clinical activity of the combination of ipilimumab (IPI) -926 in combination with cetuximab in patients with advanced head and neck cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine the dose-limiting toxicities and the recommended dose for phase 2 evaluation of the combination of IPI-926 and cetuximab in patients with advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed advanced or metastatic head and neck squamous cell (HNSCC) cancer not amenable to potentially curative resection.
* Tumor must be amenable to sequential biopsies, and patients must be willing to undergo 3 sequential tumor biopsies.
* evidence of progression after first-line chemotherapy for locally advanced or recurrent disease. There has to be at least a 4-week period since the last administration of prior therapy and initiation of the current study drugs.
* Cetuximab is indicated. However, prior therapy with cetuximab (particularly if in the primary setting) is allowed.
* Presence of measurable target on a CT-scan available for external review, with at least one diameter >/= 2cm (>/= 1cm if spiral CT-scan is used for assessment and follow-up).
* Age >/= 18 years.
* The Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >60%, see Appendix A).
* Life expectancy greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:
* leukocytes >3,000/μl
* absolute neutrophil count >1,500/μl
* platelets >100,000/μl
* total bilirubin <1.5x Upper limit normal (ULN)
* Aspartate Aminotransferase (AST)/ Alanine Aminotransferase (ALT) <2.5 X institutional upper limit of normal
* creatinine <1.5x ULN OR
* creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine above ULN.
* All women of child-bearing potential (WCBP),all sexually active male patients, and all partners of patients must agree to use adequate methods of birth control throughout the study. Women of child-bearing potential (defined as being less than 1 year post-menopausal) must have a negative serum or urine β human chorionic gonadotropin (βhCG) pregnancy test; and men and women of reproductive potential must agree to practice an effective method of avoiding pregnancy while receiving study drug and for 30 days after the final dose of study drug.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients receiving any other investigational agents.
* Patients with known brain metastases.
* History of allergic reactions attributed to cetuximab or compounds of similar chemical or biologic composition to IPI-926.
* Patients taking rifampin, St. John's wort, carbamazepine, phenytoin, and phenobarbital are excluded from this trial.
* Uncontrolled illness including, hypertension, ongoing or active infection, bleeding diathesis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Baseline Fridericia's formula (QTcF) >450 msec in men or >470 msec in women.
* Concurrent treatment with any agent known to prolong the Corrected QT (QTc) interval
* Patients who have had a venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation and meet any of the following criteria are excluded:

  * Have been on a stable dose of anticoagulation for <1 month
  * Have had a Grade 2, 3 or 4 hemorrhage in the past month
  * Are experiencing continued symptoms from their venous thromboembolic event Patients who have had a venous thromboembolic event but do not meet any of the above three criteria are eligible for participation.
* History of a seizure within the last 10 years or seizure disorder requiring anti-epileptic medications.
* Known HIV-positive patients.
* Therefore, patients taking potent inhibitors or inducers of Cytochrome P450 3A4 (CYP 3A4) should not be enrolled on this study.
* active infection or systemic use of antibiotic within 72 hours of treatment
* Cirrhotic liver disease, ongoing alcohol abuse, or chronic active or acute hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities and the recommended dose for phase 2 evaluation of the combination of IPI-926 and cetuximab | The first 3 patients enrolled will receive the first dose level. A full safety evaluation will be conducted after 6 weeks of therapy. This will continue until a MTD is determined.
  Cohorts of 3. The first cohort will receive dose level 1. A full safety evaluation will be conducted after 6 weeks. If 0/3 have a Dose limiting toxicity (DLT), then a new cohort will receive the next dose level. If 1/3 have DLT then 3 more patients will be treated at this dose level. If none has DLT then the next dose level will be administered to the next cohort; otherwise the inferior dose level will be considered the maximum tolerated dose (MTD). If 2/3 have a DLT, then the inferior dose level will be considered the MTD. In the event that the initial dose level 1 is not tolerated, a level -1 has been defined for assessment.

SECONDARY OUTCOMES:
Evaluate the clinical activity of the combination of IPI-926 with cetuximab | Patients will continue to receive treatment as long as there is evidence that their tumor is not growing and they are not experiencing any unacceptable side effects.
  Obtaining tumor biopsies at baseline, after 2 weeks of cetuximab, and after 3-4 weeks of dual therapy will enable testing our hypotheses. Patients will be assessed by standard criteria. CTs will also be conducted at the end of first cycle to assess disease progression. Confirmatory scans will also be obtained 4 weeks following initial documentation of an objective response. Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [The Journal of the National Cancer Institute (JNCI) 92(3):205-216, 2000].

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Jimeno, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States